CLINICAL TRIAL: NCT06444165
Title: Study to Assess Lebrikizumab Pen Ease of Use in Patients With Atopic Dermatitis
Brief Title: Lebrikizumab Pen Ease of Use in Participants With Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18826; J2T-MC-KGBY (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-05-31; First posted 2024-06-05 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Atopic Dermatitis
Keywords: Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lebrikizumab Pen (Experimental): Participants were instructed (following training by the study team via a training video) to simulate a single-dose subcutaneous (SC) injection using a pen by directly injecting into an injection pad. The prefilled pen contained active drug (250 milligrams (mg)/2 milliliters (mL) lebrikizumab).
  No drug was administered to the participants during this study
  Interventions: Drug: Lebrikizumab Pen

INTERVENTIONS:
Drug: Lebrikizumab Pen — Injected into a practice pad.

SUMMARY:
The purpose of this study is to assess the ease of use of the lebrikizumab pen. Participants will use a practice pad to simulate administration of a dose. Participants will complete the modified Subcutaneous Administration Assessment Questionnaire (mSQAAQ) following the simulated injection.

This study involves one study visit.

ELIGIBILITY:
Inclusion Criteria:

* Self-report being diagnosed with atopic dermatitis (AD) by a physician and able to provide approximate diagnosis date.
* Autoinjector or Pen naïve [have not used an autoinjector or pen previously; permissible to have used a pre-filled syringe (PFS) or vial and syringe].
* Willing and able to attend an in-person interview session.
* Able to complete the protocol requirements.

Exclusion Criteria:

* Cognitive or physical difficulties that could interfere with ability to understand the training, perform the injection tasks, or complete the study questionnaires as judged by the investigator.
* Are currently enrolled or have participated in the last 3 months, in a clinical study involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Is a health care practitioner who is trained in giving injections.
* Currently pregnant.
* Known hypersensitivity to any component of lebrikizumab or its excipients.
* Treatment with a live (or live attenuated) vaccine within the past 12 weeks.
* Current or chronic infection with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) per participant self-report.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 : Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Concentrics Research, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lebrikizumab Pen
Started | 55
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Lebrikizumab Pen: Participants were instructed (following training by the study team via a training video) to simulate a single-dose SC injection using a pen by directly injecting into the injection pad. The prefilled pen contained the active drug (250 mg/2 mL lebrikizumab).
  No drug was administered to the participants during this study.
Arm/Group | Lebrikizumab Pen
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.1 (16.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 54
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 30
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Responded Agree or Strongly Agree to the 'Overall Ease of Use' Question Using the Modified Subcutaneous Administration Assessment Questionnaire (mSQAAQ)
Description: mSQAAQ: This modified, short questionnaire is an instrument that includes 10 questions about the ease of use and confidence in using the lebrikizumab pen. Questions: 1) Easy for me to learn how to use, 2) Easy for me to unlock, 3) Easy to hold in my hand when I inject my dose, 4) Easy to inject my dose, 5) Easy to know that my dose is complete, 7) Easy to remove needle shield/cover, 8) Easy to pick up, 9) Overall, easy to use, 11) I am confident in my ability to use the device, and 12) I am confident my dose is complete. Responses were scored on a 7-point Likert scale ranging from 'strongly disagree' to 'strongly agree' for each question. (1) Strongly disagree; (2) Disagree; (3) Slightly disagree; (4) Neither agree nor disagree; (5) Slightly agree; (6) Agree; (7) Strongly agree. A higher score indicates greater ease and confidence in using the lebrikizumab pen.
  This endpoint reports results for Question 9: Overall, easy to use.
Time Frame: Day 1
Population: All enrolled patients
Measure: Number; unit: percentage of participants
Arm/Group | Lebrikizumab Pen
Number analyzed (Participants) | 55
percentage of participants | 96.4

2. Primary Outcome: Percentage of Participants Who Responded Agree or Strongly Agree to the ' I am Confident in my Ability to Use the Device' Question Using the mSQAAQ
Description: mSQAAQ: This modified, short questionnaire is an instrument that includes 10 questions about the ease of use and confidence in using the lebrikizumab pen. Questions 1) Easy for me to learn how to use, 2) Easy for me to unlock, 3) Easy to hold in my hand when I inject my dose, 4) Easy to inject my dose, 5) Easy to know that my dose is complete, 7) Easy to remove needle shield/cover, 8) Easy to pick up, 9) Overall easy to use, 11) I am confident in my ability to use the device, and 12) I am confident my dose is complete. Responses were scored on a 7-point Likert scale ranging from 'strongly disagree' to 'strongly agree' for each question. (1) Strongly disagree; (2) Disagree; (3) Slightly disagree; (4) Neither agree nor disagree; (5) Slightly agree; (6) Agree; (7) Strongly agree. A higher score indicates greater ease and confidence in using the lebrikizumab pen.
  This endpoint reports results for Question 11: I am confident in my ability to use the device.
Time Frame: Day 1
Population: All enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Lebrikizumab Pen
Number analyzed (Participants) | 55
percentage of participants | 96.4

ADVERSE EVENTS:
Time Frame: Baseline Up to Day 7
Description: All enrolled participants. There were no adverse events reported during this study.
Groups:
- Lebrikuzimab Pen: Participants were instructed (following training by the study team via a training video) to simulate a single-dose SC injection using a pen by directly injecting into the injection pad. The prefilled pen contained the active drug (250 mg/2 mL lebrikizumab).
  No drug was administered to the participants during this study.
Arm/Group | Lebrikuzimab Pen
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2024-04-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT06444165/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-16): https://cdn.clinicaltrials.gov/large-docs/65/NCT06444165/SAP_002.pdf